CLINICAL TRIAL: NCT06885502
Title: Personalised Health Motor and Cognitive Assistance System for RehAbilitation (PHRASE): A Randomized Clinical Trial
Brief Title: Personalised Health Motor and Cognitive Assistance System for RehAbilitation (PHRASE)
Acronym: PHRASE-2024
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eodyne Systems SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PHRASE-2024; 101058240 (Other Grant/Funding Number: Horizon Europe EIC Transition)
Record Dates: First submitted 2025-03-06; First posted 2025-03-20 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Stroke Rehabilitation; Chronic Stroke Patients; Post Stroke Recovery
Keywords: Stroke; ARAT; Motor rehabilitation; Stroke rehabilitation; Telemedicine; Virtual Reality (VR); Augmented Reality (AR); Cognitive rehabilitation; Rehabilitation at home; eHealth technology; upper limbs
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants and clinicians involved in the intervention (except those conducting the clinical assessments) will be aware of the group allocation. Outcome assessors conducting the clinical evaluations at T0 (baseline), T2 (end-intervention), and T3 (follow-up) will remain blinded to the group allocation to minimize assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (RGS) (Experimental): The standardized intervention schedule consists of daily 20-30-minute training sessions with the RGSapp, conducted at home, including weekends, for 6 weeks. This intervention is provided in addition to the prescribed conventional therapy (Standard of Care, SoC).
  Interventions: Device: RGS
- Control Group (No Intervention): The control group participants will be assessed at Baseline (T0), Week 6/End of Treatment (T2), and Follow-up at Week 14 (T3). The outcome measures will be the same as in the intervention group, including assessments of motor function, cognitive function, depression, activity participation, usability, and healthcare costs. No VR or AR-based interventions will be provided to the control group during the study period.

INTERVENTIONS:
Device: RGS — The standardized intervention schedule consists of 20-30-minute daily training sessions (including weekends) for 6 weeks, in addition to the prescribed conventional therapy (Standard of Care, SoC). Each session includes 4 to 6 exercises, each lasting approximately 5 minutes. To promote variability and engagement, at least one exercise will be replaced every week based on the participant's progress. Participants are encouraged to train more than the prescribed duration if desired. The RGSapp training will take place at home, and patients will use a smartphone. An optional wearable device (smartwatch) will be used to remotely monitor the use of the paretic upper arm for the duration of the trial. Regular check-ins by clinicians will monitor adherence, adjust the intervention if needed, and ensure the participants' safety.
  Arms: Experimental Group (RGS)

SUMMARY:
This study is a multicentric randomized controlled trial evaluating the effectiveness of digital technology, specifically a smartphone with integrated VR-and AR-based intervention, for at-home rehabilitation after stroke. The study focuses on combined motor and cognitive training for patients in the late subacute and chronic phases post-stroke. The intervention is provided through the Rehabilitation Gaming System application RGSapp, a goal-oriented, first-person virtual reality (VR) and augmented reality (AR) mobile application for upper limb rehabilitation. A total of seventy participants will be randomly assigned (1:1 ratio) to either the RGSapp intervention or conventional therapy/standard of care for six weeks. The primary outcome is motor function improvement (upper limb), assessed using the Action Research Arm Test (ARAT). Secondary outcomes include changes in cognitive function, depression, usability, adherence, validity of remote assessments, and healthcare costs.

DETAILED DESCRIPTION:
Stroke-induced motor and cognitive impairments often worsen after hospital discharge due to limited access to rehabilitation, creating a cycle of non-use and functional loss ("rehabilitation in vain"). The PHRASE system aims to counteract this by providing patient-tailored, continuous rehabilitation at home using the Rehabilitation Gaming System (RGS). This integrated approach leverages VR/AR technology, prognostic tools, and data-driven decision-making to improve motor and cognitive function, reduce costs, and enhance patient independence.

The study seeks to validate the effectiveness of the PHRASE system, focusing on its impact on motor and cognitive recovery and its use as a diagnostic and prognostic tool. It hypothesizes that combining the RGS application with conventional therapy will lead to better recovery outcomes compared to conventional therapy alone.

This randomized clinical trial (RCT) will compare the RGS-based intervention to conventional therapy in stroke patients in Spain and Romania. Participants will undergo a six-week intervention involving daily 20-30-minute RGS sessions. Assessments are at baseline, mid-study (3 weeks), end of study (6 weeks) and follow-up (14 weeks). Data will be collected on motor and cognitive function, quality of life, usability, and patient/therapist experiences.

Participants must be stroke survivors (>3 months post-stroke), aged >18, with mild to moderate upper-limb impairment (ARAT <50) and minimal smartphone experience.

The RGS-based PHRASE approach offers a scalable, cost-effective solution for continuous rehabilitation, improving patient recovery, quality of life, and reducing healthcare costs. The study aims to validate its clinical validity in real-world settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting an ischemic or intracerebral haemorrhagic stroke, ≥ 3 months post-stroke.
* Age > 18 years old
* Moderate to mild proximal upper limb motor impairment Medical Research Council Scale (MRC >2).
* ARAT: <50, inclusive, to avoid ceiling effects while allowing room for improvement.
* Able to sit on a chair or a wheelchair to interact with the RGS system.
* Minimal experience with smartphone technology based on the clinician's opinion
* Willing to participate and agree to comply with the trial scheme and procedures
* Must sign an Informed Consent Form (ICF) indicating that they understand the purpose and the procedures of the study.

Exclusion Criteria:

* Presence of a condition or abnormality that, in the opinion of the investigator, would compromise the safety of the patient or the quality of the data.
* Severe cognitive capabilities that prevent the execution of the study, evaluated by the MoCA < 19 or based on the clinician's opinion.
* Pre-stroke history of upper limb motor disability.
* Unable to use the RGS independently, according to the clinician's observations, and needing more support from a caregiver to use the RGS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Upper Limb Function (Motor Recovery) | Assessments will be conducted at Baseline (T0), End of Treatment (T2, Week 6), and Follow-up (T3, Week 14, 2-months follow-up)
  The primary objective of this study is to assess the effect of a mobile technology (RGSapp) intervention on upper limb motor function compared to Standard of Care (SoC). Upper limb function will be evaluated using the Action Research Arm Test (ARAT).
  Action Research Arm Test (ARAT) (Lyle, 1981): It is a functional assessment tool comprising 19 items, with a maximum score of 57. These items are organized into four subscales: grasp, grip, pinch, and gross movement. Each item is scored on a 4-point ordinal scale: 0 (cannot perform the task) to 3 (performs the task normally). Higher scores indicate better outcomes, reflecting greater arm function.

SECONDARY OUTCOMES:
Cognitive Function | Baseline (T0), End of Treatment (T2, Week 6), Follow-up (T3, Week 14)
  Post-stroke cognitive impairment, particularly deficits in attention, processing speed, executive function, and visual perception, which are key factors in long-term disability [Lesniak M. et al., 2008].
  Test of Attentional Performance (TAP) (Zimmermann & Fimm, 2004): It is a comprehensive battery designed to assess various aspects of attentional performance, including sustained attention, selective attention, and cognitive flexibility. It includes multiple subtests, with each scored based on accuracy and response time. Higher scores indicate better attentional capacity, providing detailed insights into different attention processes and cognitive functioning.
Depression and Mood Changes | Baseline (T0), End of Treatment (T2, Week 6), Follow-up (T3, Week 14)
  This outcome will assess depression and mood changes using the following validated tool:
  Hamilton Depression Rating Scale (HDRS) (Hamilton, 1960): It is a clinician-administered questionnaire used to evaluate the severity of depressive symptoms over the previous week, based on a structured or unstructured interview. The scale consists of 17 items, with scores ranging from 0 to 53. Higher scores indicate more severe depression, with 0-7 considered normal, 8-16 indicating mild depression, 17-23 indicating moderate depression, and 24 or above indicating severe depression.
Activity and Participation domain | Baseline (T0), End of Treatment (T2, Week 6), Follow-up (T3, Week 14)
  We will further assess the impact of stroke on parameters that strongly influence activity and participation (Activities of daily living, mobility, emotion, strength, and communication). We will use:
  Quality of Life (EQ-5D-5L) (Devlin & Brooks, 2017): It is a standardized tool for measuring health-related quality of life. It includes 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 5-point scale (1 - no problems to 5 - extreme problems). The final score is based on the combination of responses across dimensions, with higher scores reflecting better overall quality of life.
  Fatigue Severity Scale (FSS) (Krupp et al., 1988): It is a 9-item self-report questionnaire used to assess fatigue severity in individuals with chronic diseases. Each item is rated on a 1 to 7 scale, where 1 indicates no fatigue and 7 represents severe fatigue. Higher scores indicate more severe fatigue.
Usability of RGSapp | End of Treatment (T2, Week 6)
  This outcome will assess the usability of the RGSapp using the System Usability Scale (SUS).
  System Usability Scale (SUS) (Brooke, 1996): It is a 10-item questionnaire using a five-point Likert scale (Strongly Agree to Strongly Disagree) to assess the usability of products and services, including hardware, software, mobile devices, websites, and applications. Scores range from 0 to 100, with higher scores indicating better usability. A score above 68 is considered above average, below 50 suggests poor usability, and a score above 80 indicates excellent usability.
Validity of Remote Assessments Using RGSapp | Baseline (T0), End of Treatment (T2, Week 6), Follow-up (T3, Week 14)
  This outcome will assess the correlation between remote assessments using RGSapp and standard clinical evaluations of motor and cognitive function. Specifically, performance data collected through RGSapp will be compared with established clinical assessment tools, including the Action Research Arm Test (ARAT), Fugl-Meyer Assessment for Upper Extremity (FMA-UE), and Test for Attentional Performance (TAP) subtests.

CONTACTS AND LOCATIONS:
Locations (2):
- RoNeuro Institute for Neurological Research and Diagnostics, Cluj-Napoca, Romania
- Hospital Universitari Joan XXIII de Tarragona, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Only summary statistics, or disidentified datasets that pose no risk of re-identification can be shared with researchers not involved in the study to ensure transparency and reproducibility without compromising participant confidentiality.

REFERENCES:
- [Background] Cameirao MS, Badia SB, Duarte E, Frisoli A, Verschure PF. The combined impact of virtual reality neurorehabilitation and its interfaces on upper extremity functional recovery in patients with chronic stroke. Stroke. 2012 Oct;43(10):2720-8. doi: 10.1161/STROKEAHA.112.653196. Epub 2012 Aug 7. PMID 22871683
- [Background] Hidaka Y, Han CE, Wolf SL, Winstein CJ, Schweighofer N. Use it and improve it or lose it: interactions between arm function and use in humans post-stroke. PLoS Comput Biol. 2012 Feb;8(2):e1002343. doi: 10.1371/journal.pcbi.1002343. Epub 2012 Feb 16. PMID 22761551
- [Background] Ballester BR, Maier M, San Segundo Mozo RM, Castaneda V, Duff A, M J Verschure PF. Counteracting learned non-use in chronic stroke patients with reinforcement-induced movement therapy. J Neuroeng Rehabil. 2016 Aug 9;13(1):74. doi: 10.1186/s12984-016-0178-x. PMID 27506203
- [Background] Maier M, Ballester BR, Leiva Banuelos N, Duarte Oller E, Verschure PFMJ. Adaptive conjunctive cognitive training (ACCT) in virtual reality for chronic stroke patients: a randomized controlled pilot trial. J Neuroeng Rehabil. 2020 Mar 6;17(1):42. doi: 10.1186/s12984-020-0652-3. PMID 32143674